CLINICAL TRIAL: NCT04510311
Title: An Exploratory Study of 3-[18F]Fluoro-para-hydroxyphenethylguanidine ([18F]3F-PHPG) in Patients With Neuroendocrine Tumors
Brief Title: Imaging Properties of PET Radiotracer [18F]3F-PHPG in Patients With Neuroendocrine Tumors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UMCC 2019.174; HUM00167104 (Other: University of Michigan); UM-FHPG-03 (Other: University of Michigan)
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Iodine-123; 3-Iodobenzylguanidine; Positron-Emission Tomography; Tomography, X-Ray Computed; Positron Emission Tomography Computed Tomography; Tomography, Emission-Computed, Single-Photon; Single Photon Emission Computed Tomography Computed Tomography

STUDY DESIGN:
Intervention Model Description: All subjects (30 anticipated) will receive a PET/CT scan using the novel radiotracer [18F]3F-PHPG as an imaging agent. Within 60 days after the [18F]3F-PHPG PET/CT scan, approximately 12 of the subjects will also receive an FDA approved radiotracer [123I]MIBG one day prior to whole-body planar scintigraphy and SPECT/CT scans. The [123I]MIBG scans are standard clinical imaging procedures.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PET/CT scan with radiotracer [18F]3F-PHPG (Experimental): Novel radiotracer [18F]3F-PHPG prior to whole-body PET/CT scan.
  Interventions: Drug: 3-[18F]Fluoro-para-hydroxyphenethylguanidine; Diagnostic Test: Positron emission tomography/computed tomography scan
- Planar scintigraphy/SPECT scans with radiotracer [123I]MIBG (Active Comparator): FDA approved radiotracer [123I]MIBG prior to whole-body planar scintigraphy and SPECT/CT scan (standard clinical imaging procedures).
  Interventions: Drug: 3-[18F]Fluoro-para-hydroxyphenethylguanidine; Drug: [123I] metaiodobenzylguanidine; Diagnostic Test: Positron emission tomography/computed tomography scan; Diagnostic Test: Planar scintigraphy scan; Diagnostic Test: Single photon emission computed tomography/computed tomography scan

INTERVENTIONS:
Drug: 3-[18F]Fluoro-para-hydroxyphenethylguanidine — Single IV injection of 12.0 mCi (+/- 10%) [18F]3F-PHPG
  Other Names: [18F]3F-PHPG
Drug: [123I] metaiodobenzylguanidine — Single IV injection of 10.0 mCi [123I]MIBG
  Other Names: [123I]MIBG; AdreView™
  Arms: Planar scintigraphy/SPECT scans with radiotracer [123I]MIBG
Diagnostic Test: Positron emission tomography/computed tomography scan — Whole-body PET/CT scan performed at two time-points: 1.5 hours and 3 hours after IV injection of [18F]3F-PHPG
  Other Names: PET/CT
Diagnostic Test: Planar scintigraphy scan — Whole-body scan using planar scintigraphy with a gamma camera performed the day after IV injection of [123I]MIBG
  Arms: Planar scintigraphy/SPECT scans with radiotracer [123I]MIBG
Diagnostic Test: Single photon emission computed tomography/computed tomography scan — SPECT/CT scan of the primary neuroendocrine tumor performed the day after IV injection of [123I]MIBG
  Other Names: SPECT/CT scan
  Arms: Planar scintigraphy/SPECT scans with radiotracer [123I]MIBG

SUMMARY:
The goal of this exploratory study is to test whether [18F]3F-PHPG can be used reliably to map the locations of tumors in patients with neuroendocrine tumors. If so, the results of this study will be used to support further development of [18F]3F-PHPG as a clinical tool for neuroendocrine tumor localization and staging.

DETAILED DESCRIPTION:
Subjects enrolled in this study will be recruited from the population of adult patients with neuroendocrine tumors, including pheochromocytoma and paraganglioma, being treated at the University of Michigan Hospital.

The primary objective of the study is to obtain basic information on the biodistribution and pharmacokinetics of [18F]3F-PHPG in cancer patients with neuroendocrine tumors.

The secondary objective of the study is to compare the diagnostic performance of [18F]3F-PHPG in cancer patients with neuroendocrine tumors with the FDA approved radiopharmaceuticals [123I]metaiodobenzylguanidine ([123I]MIBG) and [68Ga]DOTA-TATE in the same patients. A group of approximately 12 of the subjects scanned with [18F]3F-PHPG will be recruited to undergo a whole-body [123I]MIBG scan using planar scintigraphy with a gamma camera, following the standard clinical protocol used at the University of Michigan. In addition, a single SPECT/CT scan of the primary neuroendocrine tumor will be acquired after the whole-body scan to provide a tomographic image for comparison with the positron emission tomography (PET) image acquired using [18F]3F-PHPG. Several subjects enrolled on this study will undergo [68Ga]DOTA-TATE scans off-study, as part of routine clinical management. Existing [68Ga]DOTA-TATE scans will be obtained from consenting subjects' medical records.

This is an exploratory study and thus all statistical data analyses will be exploratory in nature.

ELIGIBILITY:
Inclusion Criteria:

* Current neuroendocrine tumor diagnosis
* Able to lie flat for 60 minutes
* Provision of informed consent

Exclusion Criteria:

* Pregnancy or lactation
* Claustrophobia
* Inability to lie flat for 60 minutes
* Currently taking medications that may alter PET scans of neuroendocrine tumors with these tracers, including any of the following:

  * Tricyclic antidepressants, which inhibit the norepinephrine transporter: desipramine, amitriptyline, imipramine
  * Cold medications containing the sympathomimetic amines: phenylephrine, phenylpropanolamine, pseudoephedrine
  * Nasal decongestants (some use phenylephrine as the active agent)
  * Cocaine (which inhibits the norepinephrine transporter)
  * Tetrabenazine (Xenazine), which inhibits the VMAT2 transporter
  * Monoamine oxidase inhibitors (MAOI)
  * Some antihypertensive drugs: reserpine, labetalol, α-methyldopa, clonidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Image quality assessed by standardized uptake values | Up to 180 minutes
  The maximum standardized uptake value (SUVmax) of [18F]3F-PHPG in neoplastic lesions will be quantified from the PET images using region-of-interest (ROI) analysis.
Biodistribution of [18F]3F-PHPG | 90 minutes and 180 minutes after administration of tracer
  Changes in the measured tissue concentrations (kBq/cc) of [18F]3F-PHPG in neoplastic lesions and abdominal organs from the two acquired PET images (acquired at 90 min and 180 min after tracer injection).

CONTACTS AND LOCATIONS:
Overall Officials: David Raffel, Ph.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No